CLINICAL TRIAL: NCT04072692
Title: Investigation of the Relation Between Trigger Digit and Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A-ER-103-404
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: The Comorbidity Between the Trigger Digit and Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1st part: The gliding properties of the tendons (No Intervention): No intervention. Subjects are measured by ultrasound under 5 different postures of the hand for forty minutes.
- 1st part: The gliding properties of the median nerve (No Intervention): No intervention. Subjects are measured by ultrasound under under 6 different postures of the wrist and hand and 5 different movement patterns of the wrist and hand for forty minutes.
- 2nd part: New hybrid rehabilitation strategy (Experimental): The program includes pre-test, 8 times training, post-test and follow-up test.
  For pre-test, subjects perform the specific hand movement under different exerting force conditions and 4 different angles of phalangeal joints and be asked to do Phalen test, Grip strength test, Pinch test and SWMT test. It takes 40 minutes.
  For post-test, the same procedure is repeated again after completing all training.
  For follow-up, the same procedure is repeated again 6 months after completing all training.
  After pre-test, 8 times hybrid rehabilitation training are asked. There are two times in a week, and all training will be completed in one month. Each time will take forty minutes.
  Interventions: Other: Hybrid rehabilitation training
- 2nd part: Traditional strategy (Experimental): The program includes pre-test, 8 times training, post-test and follow-up test.
  For pre-test, subjects perform the specific hand movement under different exerting force conditions and 4 different angles of phalangeal joints and be asked to do Phalen test, Grip strength test, Pinch test and SWMT test. It takes 40 minutes.
  For post-test, the same procedure is repeated again after completing all training.
  For follow-up, the same procedure is repeated again 6 months after completing all training.
  After pre-test, 8 times traditional rehabilitation training are asked. There are two times in a week, and all training will be completed in one month. Each time will take forty minutes.
  Interventions: Other: Traditional rehabilitation training
- 3rd part: The effect of carpal tunnel release (No Intervention): No intervention. The program includes pre-test, post-test and two times follow-up tests.
  For pre-test, subjects perform the mechanical properties of the flexor tendon assessment and functional assessment of both hands before carpal tunnel release surgery. It takes 40 minutes.
  For post-test, subjects perform the functional assessment of both hands one week after carpal tunnel release surgery. It takes 20 minutes.
  For first follow-up, subjects perform the mechanical properties of the flexor tendon assessment and functional assessment of both hands one month after carpal tunnel release surgery. It takes 40 minutes.
  For second follow-up, subjects perform the mechanical properties of the flexor tendon assessment and functional assessment of both hands two month after carpal tunnel release surgery. It takes 40 minutes.
- 3rd part: Wearable anti-bowstringing orthosis (WABO) (Experimental): The program includes pre-test, post-test and two times follow-up tests.
  For pre-test, subjects perform the mechanical properties of the flexor tendon assessment and functional assessment of both hands before carpal tunnel release surgery. It takes 40 minutes.
  Subjects wear WABO in the morning and a splint at night within a week after carpal tunnel release surgery.
  For post-test, subjects perform the functional assessment of both hands with and without wearing WABO and a splint one week after carpal tunnel release surgery. It takes 40 minutes.
  From the third weeks after carpal tunnel release surgery, subjects wear WABO only in the morning.
  For first follow-up, the same procedure in pre-test is repeated again one month after carpal tunnel release surgery. It takes 40 minutes.
  For second follow-up, the same procedure in pre-test is repeated again two month after carpal tunnel release surgery.
  Interventions: Other: Wearable anti-bowstringing orthosis (WABO)

INTERVENTIONS:
Other: Hybrid rehabilitation training — Hybrid rehabilitation training is modified tendon gliding exercise with median nerve mobilization.
  Arms: 2nd part: New hybrid rehabilitation strategy
Other: Traditional rehabilitation training — Traditional rehabilitation training uses traditional physiotherapy, such as splint, therapeutic ultrasound and electrotherapy.
  Arms: 2nd part: Traditional strategy
Other: Wearable anti-bowstringing orthosis (WABO) — WABO is a custom-designed orthosis to restrict the bowstringing effect of the flexor tendon in the carpal tunnel.
  Arms: 3rd part: Wearable anti-bowstringing orthosis (WABO)

SUMMARY:
The purpose of this study is to comprehend the association between the trigger digit and carpal tunnel syndrome based on the quantification of the tendon and nerve characteristics. It includes three parts.

The first part is an observational study. The aim of the first part is to attempts to measure the gliding and morphological characteristics of the flexor tendons and median nerve in the longitudinal or cross-sectional directions via the ultrasonographical images incorporating with the motion capture experiment of the wrist and fingers. The gliding and morphological features of the tendons and nerve will be compared under different postures or movement patterns of the wrist and hand.

The second part is an interventional study. The aim of the first part is to establishes a novel hybrid rehabilitation protocol which combines the tendon gliding exercise with nerve mobilization to treat either the trigger digit or the carpal tunnel syndrome. A randomized controlled trial to investigate the short-term treatment effect and the follow-up examination will be carried out as well.

The third part is an observational study. The aim of the first part is to investigate the effects of carpal tunnel release on the hand performances from functional perspectives. In addition, a novel wrist orthosis will be developed to eliminate the bowstringing effect of the flexor tendons after carpal tunnel release.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects without any history musculoskeletal diseases
2. Patients with carpal tunnel release surgery

Exclusion Criteria:

* Subjects with fracture or surgery in the upper extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Change in the gliding features of tendons | baseline, 1 month, 6 months
  The gliding features of tendons is measured by ultrasound images of the flexor tendons
Change in the gliding features of median nerve | baseline, 1 month, 6 months
  The gliding features of median nerve is measured by ultrasound images of the flexor tendons
Change in the grip strength | baseline, 1 month, 6 months
  Grip strength is measured by a grip strength meter.
Change in the pinch force | baseline, 1 month, 6 months
  Three types of pinch force are measured by a pinch gauge.
Change in the threshold value of sensitivity | baseline, 1 month, 6 months
  Threshold value of sensitivity is examined by using Semmes-Weinstein Monofilament testing.
Change in the mechanical properties of the flexor tendons | baseline, 1 month, 6 months
  The mechanical properties are examined by measuring torque value contributed by the flexor tendons and movements of the flexor tendons

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan